CLINICAL TRIAL: NCT02907281
Title: A 3-year, Multi-center Study to Evaluate Optical Coherence Tomography as an Outcome Measure in Patients With Multiple Sclerosis
Brief Title: Optical Coherence Tomography (OCT) Trial in Multiple Sclerosis
Acronym: OCTIMS
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CFTY720D2319; 2011-001437-16 (EudraCT Number)
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Multiple Sclerosis; RRMS
Keywords: Multiple sclerosis,; MS,; Optical coherence tomography; OCT,; RRMS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Multiple sclerosis patients: Multiple sclerosis patients
  Interventions: Other: Observational
- Healthy volunteers: Healthy volunteers
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
This is a 3-year, pharmacologically non-interventional study to evaluate OCT as an outcome measure in patients with relapsing remitting multiple sclerosis (RRMS).

Approximately 350 RRMS patients, either untreated or treated with an approved MS disease-modifying therapy and approximately 70 reference subjects without ophthalmologic or neurologic disease are enrolled. No study medications are provided. Patients on disease-modifying therapy are treated according to the local prescribing information. For each MS patient and each reference subject, the study consists of Screening (up to 1 month), Baseline, and a 36-month longitudinal data collection phase. Eligibility will be confirmed during Screening.

ELIGIBILITY:
Multiple sclerosis patients

* A diagnosis of MS as defined by the 2005 revision to the McDonald criteria with a relapsing-remitting course
* MS disease duration of more than one year (from diagnosis of MS) before study entry

Healthy volunteers

- Matched to MS patients based on age, gender, ethnicity and visual refraction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Sclerosis patients and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2012-05-29 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
Change in Retinal Nerve Fiber Layer Thickness (RNFL) | 36 months
  evaluate change in RNFL thickness in relapsing remitting multiple sclerosis (RRMS) patients followed for up to 36 months compared to a group of reference subjects (without neurologic or ophthalmic disease) to determine whether the technology is sufficiently sensitive to disease and to change over time.

SECONDARY OUTCOMES:
Correlation of change in macular volume with change in brain volume | 36 months
  To evaluate the correlation of change in macular volume with change in brain volume as measured by MRI in RRMS patients followed for up to 36 months.
Assess reproducibility of RNFL thickness on optical coherence tomography | 4 weeks
  To evaluate short-team reproducibility of the RNFL thickness measure at study start by test/re-test estimation after a 4-week interval in RRMS patients and reference subjects (without neurologic or ophthalmic disease).
Change in macular volume over 36 months | 36 months
  To evaluate change in macular volume over 36 months in RRMS patients compared to a group of reference subjects (without neurologic or ophthalmic disease).
Correlation of change in RNFL thickness with change in brain volume | 36 months
  To evaluate the correlation of change in RNFL thickness with change in brain volume as measured by magnetic resonance imaging (MRI) in RRMS patients followed for up to 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- United States (5):
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Iowa City, Iowa
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Philadelphia, Pennsylvania
- Australia (2):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Parkville, Victoria
- Canada (2):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Greenfield Park, Quebec
- Novartis Investigative Site, Prague, Czechia
- Novartis Investigative Site, Copenhagen, Denmark
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Magdeburg
- Italy (7):
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Bari
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Montichiari
  - Novartis Investigative Site, Padua
  - Novartis Investigative Site, Roma
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Lodz, Lódzkie, Poland
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Zurich, Switzerland
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes